CLINICAL TRIAL: NCT02058017
Title: The Signal Transducer and Activator of Transcription (STAT)3 Pathway and the Development of STAT3 Phosphorylation Inhibitors as Cancer Therapy: Lead-In Phase I Dose-Escalating, Open-Label, Non-Randomised Study of A Weekly Regimen OPB-51602 in Advanced Refractory Solid Tumours With Enrichment Cohorts of Nasopharyngeal Carcinoma Followed By A Biomarker Study Evaluating OPB-51602 in Locally Advanced Nasopharyngeal Carcinoma Prior to Definitive Chemoradiotherapy
Brief Title: OPB-51602 in Locally Advanced Nasopharyngeal Carcinoma Prior to Definitive Chemoradiotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lactic and metabolic acidosis of OPB-51602 is not tolerable
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry); Shin Nippon Biomedical Laboratories, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP01/27/13; 2013/00691 (Other: NHG Domain Specific Review Board)
Record Dates: First submitted 2014-01-15; First posted 2014-02-07 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Part I & Part II (Experimental): Part I - This is a lead-in dose-finding, open-label, non-randomised arm of the study: Using a starting dose of 10mg per week, an accelerated dose titration escalation followed by a 3+3 design will be employed until MTD and recommended weekly dose are determined.
  Part II - This is a single-centre, open-label non-randomised phase II study evaluating OPB-51602 in stage III-IVB NPC conducted in the window period prior to definitive chemoradiotherapy. Eligible patients will receive OPB-51602 on a weekly basis (Day 1, 8, 15) at the recommended dose determined in part I for a total of 15 days prior to definitive chemoradiotherapy.
  Interventions: Drug: OPB-51602

INTERVENTIONS:
Drug: OPB-51602
  Other Names: OPB-51602 OPB-51602 is an inhibitor of STAT3 phosphorylation developed by Otsuka Pharmaceuticals, Japan.

SUMMARY:
This is a lead-in dose escalation study to determine the safety, tolerability, pharmacokinetics, maximum tolerated dose (MTD), and recommended Phase II dose of OPB-51602 administered on a weekly basis in subjects with advanced malignancies. Using the recommended phase II dose, the efficacy and tolerability of OPB-51602 administered prior to definitive chemoradiotherapy will be evaluated in locally advanced NPC patients. This study's overarching goal is the development of STAT3 inhibitors as a novel class of anti-cancer agents and the optimization of patient selection for STAT3 inhibitor therapy through parallel biomarker studies. This study hopes to establish a therapeutic window for OPB-51602 in solid tumours and will evaluate its potential as a targeted therapy of NPC, since this represents a critical unmet clinical need. The development of predictive and pharmacodynamic biomarkers in tandem with the clinical evaluation of OPB-51602 will be crucial to its therapeutic advancement and will enable an understanding of the genetic contexts of responsiveness and resistance to OPB-51602, which can in turn lead to the development of effective drug combinations to overcome resistance.The study hypothesizes that OPB-51602, a first-in-class STAT3 inhibitor, is efficacious in solid tumours with constitutively activated STAT3, such as NPC.

DETAILED DESCRIPTION:
Part I This is a lead-in dose-finding, open-label, non-randomised study of OPB-51602 in patients with advanced refractory solid tumours who have biopsy-amenable lesions at study entry. Using a starting dose of 10mg per week, an accelerated dose titration escalation followed by a 3+3 design will be employed until MTD and recommended weekly dose are determined. Following this, an expansion cohort of 10 patients will be enrolled to establish safety of the recommended phase II dose. Additionally, it is also planned to explore the efficacy of the agent in an enrichment cohort of approximately 10 metastatic NPC patients. One treatment cycle is defined as a period of 28 days. Tumour biopsies will be performed at baseline while blood sampling for circulating biomarkers will be performed on days 1, 2, 3, 8, 22 and upon completion of OPB-51602 dosing. Pharmacokinetic sampling will be done on Cycle 1 Days 1, 8 and 22. Safety assessments will be performed weekly till week 8, bi-weekly till week 16, then monthly thereafter and response assessments will be performed every 8 weeks. The number of subjects estimated to participate in this study will depend on the number of cohorts enrolled.

Part II This is a single-centre, open-label non-randomised phase II study evaluating OPB-51602 in stage III-IVB NPC conducted in the window period prior to definitive chemoradiotherapy. Eligible patients will receive OPB-51602 on a weekly basis (Day 1, 8, 15) at the recommended dose determined in part I for a total of 15 days prior to definitive chemoradiotherapy. Response assessment will be performed after OPB-51602 dosing on day 15 using PET/CT scans and clinical tumour measurements, while other radiologic assessments will be performed on the completion of chemoradiotherapy. Safety assessments will be performed at weekly intervals until day 22 or until toxicities related to the study treatment have been resolved. Tumour biopsies will be performed at baseline and day 15 while circulating biomarker studies will be performed on days 1, 2, 3, 8, 15 and upon completion of chemoradiotherapy. There is no mandated rest period between the administration of study drug and definitive chemoradiotherapy. The decision to proceed with chemoradiotherapy is at the discretion of individual investigators, provided the subject has recovered or is recovering from all significant toxicities of the study drug. Chemoradiotherapy should be in accordance with the institutional standard and induction chemotherapy is not permitted. Proposed alternative treatment regimens must receive the approval of the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Part I only: Patients with pathologically confirmed, locally recurrent or metastatic solid tumours who have failed standard treatment options. In the enrichment cohort, NPC patients will be eligible as long as they have received prior platinum-based therapy, either in the curative or metastatic setting. At least one tumour lesion (primary or metastatic) that is suitable for baseline biopsy which is accessible either by free hand or image guided biopsy is required.
* Part II only: Patients with histologically confirmed WHO Type III NPC. Tumour stage III, IVA (T4 N0-2 M0) or IVB (Any T N3 M0) according to the American Joint Committee on Cancer (AJCC) 2010 criteria and planned for definitive chemoradiotherapy (radiotherapy at 70Gy/33# with concurrent IV cisplatin 40mg/m2/week for duration of radiotherapy) as per institutional standards. Patients who are planned for induction chemotherapy followed by concurrent chemoradiotherapy will not be included in the study. Patients receiving alternative chemoradiotherapy regimens may only be considered upon approval of the P.I.
* Age ≥ 21 years at the time of consent
* Eastern Cooperative Oncology Group (ECOG) performance status < 1
* Life expectancy > 3 months
* Adequate organ function as defined by:

Bone marrow function

* Haemoglobin ≥ 9g/dl
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 75 x 109/L. Liver function
* Bilirubin </= 2.5x upper limit of normal (ULN)
* Alanine transaminase (ALT) and aspartate transaminase (AST) </= 2.5x ULN or </= 5x ULN if liver metastases are present
* Prothrombin time (PT) within the normal range for the institution. Renal function
* Plasma creatinine </=1.5x institutional ULN for part I and calculated creatinine clearance (by the Cockcroft-Gault formula) > 60mL/min for part II.
* Capable of swallowing OPB-51602 tablets
* Recovery from any previous drug- or procedure-related toxicity to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 Grade 0 or 1 (except alopecia), or to baseline preceding the prior treatment.
* Signed informed consent obtained before any study specific procedure. Subjects must be able to understand and be willing to sign the written informed consent.

Exclusion Criteria:

* Part I only: Chemotherapy, radiotherapy, surgery, immunotherapy or other therapy within 4 weeks of starting investigational medicinal product (IMP).
* Part II only: Previous or concurrent anti-cancer chemotherapy, immunotherapy, radiotherapy or any other investigational therapy.
* Uncontrolled central nervous system metastasis (applicable to Part I)
* Any concomitant condition that could compromise the objectives of this study and/or the patient's compliance (eg. severe medical conditions such as uncontrolled infection, poorly controlled diabetes mellitus, hypercalcaemia, psychiatric disorders).
* Use of any of the prohibited medications and other substances listed in Appendix 2 (CYP3A4 Inhibitors and Inducers) within 1 week prior to start of study drug administration
* Pregnancy or breastfeeding.
* Women of childbearing potential not employing adequate contraception. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of study medication, and a negative result must be documented before start of study medication. Women of childbearing potential and men, must agree to use adequate contraception (barrier method of birth control) upon signing the informed consent form until at least 3 months after the last study drug administration.
* Known or suspected allergy to the investigational agent or any agent given in association with this study.
* Previous or concurrent cancer which is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumours (Ta, Tis & T1) or any cancer curatively treated > 3 years prior to study entry.
* Interstitial lung disease with ongoing signs and symptoms at the time of screening.
* Patients with CTCAE Grade 2 or higher peripheral neuropathy.
* Patients with CTCAE Grade 1 or higher pneumonitis (interstitial pneumonia) or pulmonary fibrosis
* History of significant cardiac disease: congestive cardiac failure > NYHA class II, ongoing unstable angina, new-onset angina or myocardial infarction within the past 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Recommended Phase II dose of OPB-51602 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wong, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore